CLINICAL TRIAL: NCT07367620
Title: Immediate Mechanical Complications After Central Venous Catheterization; a Multicentre Cohort Study
Brief Title: Immediate Mechanical Complications After Central Venous Catheterization
Acronym: CATH-RISK
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Kander (Other)
Collaborators: Region Skane (Other); Lund University (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Professor, Region Skane
Organization: Region Skane (Other)
Other Study IDs: CATH-RISK
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Central Venous Access Complications
Keywords: central venous catheters; Catheterization, Central Venous; Vascular Access Devices
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing central venous catheterization: This cohort includes adolescent and adult patients undergoing central venous catheter insertion as part of routine clinical care at participating hospitals. Catheterizations are performed according to local clinical guidelines and standard practice, predominantly using real-time ultrasound guidance. No study-specific interventions are mandated.
  Data on patient characteristics, operator factors, procedural details, and immediate mechanical complications occurring after catheter insertion are collected from existing electronic health record-based registries. The study is purely observational and does not influence clinical decision-making, choice of catheterization technique, or patient management.
  Interventions: Device: Central Venous Catheterization

INTERVENTIONS:
Device: Central Venous Catheterization — No intervention is assigned in this study. Central venous catheter insertions are performed according to standard clinical practice and local guidelines at participating hospitals. The study involves observational data collection only, using information routinely documented in the electronic health record and clinical registries. No changes to patient management, catheterization technique, or follow-up are introduced as part of the study.

SUMMARY:
The goal of this observational study is to determine the incidence of immediate mechanical complications after central venous catheterization and to explore factors associated with major mechanical complications in adolescent and adult patients undergoing central venous catheter insertion in routine clinical care.

The main questions it aims to answer are:

What is the incidence of immediate mechanical complications, including major complications, following central venous catheterization?

Which patient-, operator-, and procedure-related factors are associated with major mechanical complications?

To what extent can these factors be combined to estimate the risk of major mechanical complications before catheter insertion?

This study builds on a previous multicentre registry study of central venous catheterization but includes a substantially larger number of catheter insertions. An additional exploratory objective is to assess the feasibility of developing a risk estimation model (CATH-RISK) for major mechanical complications based on available data.

Participants will have their central venous catheter insertions and related clinical data recorded in an existing clinical registry. No interventions beyond standard clinical care will be performed.

DETAILED DESCRIPTION:
Central venous catheterization is a common invasive procedure in anaesthesia, intensive care, and emergency medicine, but it is associated with a risk of immediate mechanical complications ranging from minor events to rare but potentially life-threatening major complications. Although the widespread use of real-time ultrasound guidance has reduced complication rates, major mechanical complications continue to occur and remain clinically important.

This observational registry study (CATH-RISK) is designed to extend a previously conducted multicentre cohort study of mechanical complications after central venous catheterization by substantially increasing the number of included catheter insertions. The larger dataset will allow more precise estimation of complication rates and more robust assessment of factors associated with major mechanical complications occurring in close temporal relation to catheter insertion.

All central venous catheter insertions performed in participating hospitals during the study period will be identified through existing electronic health record-based registries. Mechanical complications occurring within a predefined time window after catheter insertion will be systematically recorded and classified according to predefined criteria. Patient-related, operator-related, and procedure-related variables routinely available in clinical documentation will be extracted for analysis.

The primary objective of the study is to determine the incidence of immediate mechanical complications, including major mechanical complications, after central venous catheterization in contemporary clinical practice. Secondary objectives include identifying factors associated with major mechanical complications and describing their relative contributions.

An additional exploratory objective is to assess the feasibility of combining selected variables into a risk estimation model (CATH-RISK) for major mechanical complications. Given the expected low incidence of major complications, any modelling will be considered hypothesis-generating and aimed at evaluating potential clinical usefulness rather than establishing a definitive prediction tool.

The study is purely observational and does not involve any deviation from standard clinical care. No study-specific interventions will be performed, and no additional procedures, examinations, or follow-up visits will be required for participants.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a central venous catheter within the study period will be observed

Exclusion Criteria:

* Patients who die within 24 hours for reasons unrelated to the catheterization will be excluded, whereas patients whose death is directly related to the central venous catheterization will be included

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving a central venous catheter within the study period will be observed
Sampling Method: Non-Probability Sample
Enrollment: 29500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Number of cases with bleeding grade 3-4 | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Grade 3 bleedings/hematoma formation/hemothorax (bleedings requiring invasive intervention or blood transfusion) or arterial catheter placement and grade 4 bleedings/hemothorax (life-threatening bleedings). All grade 3-4 bleedings will be classified as major mechanical complications.
Number of cases with arrhythmia grad 3-4 during the inserting procedure | During the procedure of inserting the central venous catheter
  Mechanical complication during the CVC-insertion. Recognized at the continuous ECG by the inserting physician or the assistant. Arrhythmias grade 3 (symptomatic arrhythmia requiring urgent medical intervention) and grade 4 (symptomatic arrhythmia with life-threatening consequences) will be considered major mechanical complications.
Number of cases with pneumothorax at post-procedural x-ray of the thorax | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Pneumothoraces will be detected using x-ray after the central venous catheter insertion. All pneumothoraces will be classified as major mechanical complications
Number of cases with persistent nerve injury classified as sensory loss, paraesthesia or loss of motor neuron function | Persistent more than 72 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected and documented by the patient responsible physician or nurse. Will be considered a major mechanical complication.

SECONDARY OUTCOMES:
Number of cases with failure to place the catheter | During the procedure of inserting the central venous catheter
  An attempt to insert a central venous catheter was performed but failed. Will be detected by the inserting anesthesiologist. Will be classified as minor mechanical complications.
Number of cases with bleeding grad 2 | Up to 24 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Grade 2 bleedings/hematoma formation (bleedings requiring external compression) or arterial puncture with the steel canula. Will be detected during the inserting procedure or at the daily inspection by the patient responsible physician or nurse. Will be considered minor mechanical complications.
Number of cases with arrhythmia grad 1-2 during the inserting procedure | During the procedure of inserting the central venous catheter
  Mechanical complication during the CVC-insertion. Recognized at the continuous ECG by the inserting physician or the assistant. Arrhythmias grade 1 (asymptomatic arrhythmia not requiring intervention) and grade 2 (asymptomatic or symptomatic arrhythmia requiring non-urgent medical intervention) will be considered minor mechanical complications.
Number of cases with transient nerve injury classified as sensory loss, paraesthesia or loss of motor neuron function | Transient up to 72 hours after insertion of the central venous catheter
  Mechanical complication after CVC-insertion. Will be detected and documented by the patient responsible nurse. Will be considered a minor mechanical complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected in this study will not be made publicly available. De-identified data may be shared with qualified researchers upon reasonable request, subject to approval by the study steering committee and applicable ethical and legal regulations. Requests should include a methodologically sound research proposal and may require a data use agreement.
Supporting Information: CSR
Time Frame: Data will be available beginning after publication of the primary study results, with no defined end date
Access Criteria: De-identified individual participant data may be shared with qualified researchers upon reasonable request and approval by PI, in accordance with ethical and data protection regulations. Data will be shared via secure transfer after execution of a data use agreement